CLINICAL TRIAL: NCT00485732
Title: A Phase IIIb, Double-blind, Randomized, Controlled Study to Evaluate the Immunogenicity and Safety of GlaxoSmithKline Biologicals' HPV-16/18 L1 VLP AS04 Vaccine, Administered Intramuscularly in Healthy Female Subjects Aged 15 - 25 Years
Brief Title: A Study to Evaluate the Immune Response and Safety of GSK Biologicals' HPV-16/18 L1 VLP AS04 Vaccine/Cervarix TM Vaccine in Healthy Females Aged 15-25 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 107291
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Results first posted 2009-12-17 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2016-11

CONDITIONS: Infections, Papillomavirus
Keywords: Cervical neoplasia; AS04; Randomized; Cervical cancer; HPV-16/18 L1 VLP AS04; Phase IIIb; Korea; HPV; Double-blind; Controlled
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Cervarix Group (Experimental)
  Interventions: Biological: HPV-16/18 VLP/AS04 vaccine (Cervarix TM)
- Placebo Group (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: HPV-16/18 VLP/AS04 vaccine (Cervarix TM) — Three doses of vaccine administered intramuscularly according to a 0, 1, 6-month schedule.
  Other Names: GSK Biologicals' HPV-16/18 VLP/AS04 vaccine
  Arms: Cervarix Group
Biological: Placebo — Three doses of placebo administered intramuscularly according to a 0, 1, 6-month schedule.
  Arms: Placebo Group

SUMMARY:
Human papillomavirus infection has clearly been recognized as the cause of cervical cancer. The infection of the cervix by certain oncogenic types of HPV, if not cleared, can lead to cervical cancer in women. This study will evaluate the immunogenicity and safety of the GSK Biologicals' HPV-16/18 L1 VLP AS04 vaccine (Cervarix TM) vaccine.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they or their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* A female between, and including, 15 and 25 years of age at the time of the first vaccination.
* Written informed assent obtained from the subject and informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects must have a negative urine pregnancy test.
* Subjects of childbearing potential at the time of study entry must be abstinent, or must be using adequate contraceptive precautions for 30 days prior to vaccination and must agree to continue such precautions for two months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study/ control vaccine within 30 days preceding the first dose of study/ control vaccine, or planned use during the study period.
* Pregnant or breastfeeding.
* Planning to become pregnant or likely to become pregnant.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after the first dose of vaccine. However, the administration of routine vaccines up to 8 days before the first dose of study vaccine is allowed. Enrolment will be deferred until the subject is outside of specified window.
* Previous administration of components of the investigational vaccine
* Previous vaccination against HPV or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period.
* Any medically diagnosed or suspected immunodeficient condition such as HIV infection based on medical history and physical examination.
* History of thrombocytopenia or hemostatic disorder in which case the study vaccine should under no circumstances be administered intramuscularly.
* History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the study/control vaccines.
* Hypersensitivity to latex.
* Known acute or chronic, clinically significant neurologic, pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by previous physical examination or laboratory tests.
* History of chronic condition(s) requiring treatment.
* Administration of immunoglobulins and/or any blood product within three months preceding the first dose of study/control vaccine or planned administration during the study period. Enrolment will be deferred until the subject is outside of specified window.
* Acute disease at the time of enrolment.

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 225 (Actual)
Dates: Start 2007-06-11; Primary Completion 2008-03-30 (Actual); Study Completion 2008-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Kim SC, Song YS, Kim YT, Kim YT, Ryu KS, Gunapalaiah B, Bi D, Bock HL, Park JS. Human papillomavirus 16/18 AS04-adjuvanted cervical cancer vaccine: immunogenicity and safety in 15-25 years old healthy Korean women. J Gynecol Oncol. 2011 Jun 30;22(2):67-75. doi: 10.3802/jgo.2011.22.2.67. PMID 21860731
- [Background] Verstraeten T, Descamps D, David MP, Zahaf T, Hardt K, Izurieta P, Dubin G, Breuer T. Analysis of adverse events of potential autoimmune aetiology in a large integrated safety database of AS04 adjuvanted vaccines. Vaccine. 2008 Dec 2;26(51):6630-8. doi: 10.1016/j.vaccine.2008.09.049. PMID 18845199
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 107291 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107291 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107291 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107291 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107291 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 107291 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107291 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Cervarix Group: Subjects received 3 doses of HPV-16/18 VLP/AS04 vaccine (Cervarix TM) vaccine administered intramuscularly according to a 0, 1, 6-month schedule.
- Placebo Group: Subjects received 3 doses of placebo according to a 0, 1, 6-month schedule.
Period: Overall Study
Arm/Group | Cervarix Group | Placebo Group
Started | 149 | 76
Completed | 141 | 67
Not Completed | 8 | 9
Not completed — Protocol Violation | 1 | 3
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix Group | Placebo Group | Total
Number analyzed (Participants) | 149 | 76 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.0 (2.24) | 21.9 (2.63) | 22.0 (2.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 76 | 225
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Seroconverted for Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibodies
Description: Seroconversion is defined as the appearance of anti-HPV-16 and/or anti-HPV-18 antibodies (i.e. antibody titer ≥ cut-off value) in the sera of subjects seronegative before vaccination.
  Cut-off values were 8 enzyme-linked immunosorbent assay units per milliliter (EL.U/mL) for anti-HPV-16 antibodies and 7 EL.U/mL for anti-HPV-18 antibodies.
Time Frame: One month post Dose 3 (Month 7)
Population: Analysis was performed on initially seronegative subjects from the According-to-Protocol (ATP) cohort for immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 125 | 61
Participants
  Anti-HPV-16 | 125 | 2
  Anti-HPV-18: number analyzed (Participants) | 122 | 60
  Anti-HPV-18 | 122 | 3

2. Secondary Outcome: Anti-HPV-16 and Anti-HPV-18 Antibody Titres
Description: Titres are given as geometric mean titres (GMTs) calculated on all subjects.
Time Frame: Before vaccination (PRE) and one month post Dose 3 (Month 7)
Population: Analysis was performed on the ATP cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: titre
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 136 | 67
titre
  Anti-HPV-16 (PRE) | 4.6 [4.2 to 5.1] | 4.8 [4.1 to 5.7]
  Anti-HPV-16 (Month 7) | 9226.4 [8085.4 to 10528.4] | 4.9 [4.2 to 5.8]
  Anti-HPV-18 (PRE): number analyzed (Participants) | 135 | 67
  Anti-HPV-18 (PRE) | 4.1 [3.7 to 4.4] | 4.0 [3.5 to 4.5]
  Anti-HPV-18 (Month 7): number analyzed (Participants) | 135 | 66
  Anti-HPV-18 (Month 7) | 4240.2 [3692.1 to 4869.7] | 4.3 [3.7 to 5.0]

3. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling at the injection site.
Time Frame: During the 7-day (Days 0-6) period following each vaccination
Population: Analysis was performed on the Total vaccinated cohort on the subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 145 | 72
Participants
  Pain | 140 | 64
  Redness | 109 | 35
  Swelling | 89 | 19

4. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed include arthralgia, fatigue, fever, gastrointestinal symptoms, headache, myalgia, rash, and urticaria.
Time Frame: During the 7-day (Days 0-6) period following each vaccination
Population: Analysis was performed on the Total vaccinated cohort on the subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 145 | 72
Participants
  Arthralgia | 35 | 8
  Fatigue | 103 | 39
  Fever | 7 | 2
  Gastrointestinal symptoms | 52 | 16
  Headache | 73 | 30
  Myalgia | 97 | 33
  Rash | 29 | 8
  Urticaria | 12 | 2

5. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AE)
Description: Unsolicited adverse event= Any adverse event (AE) reported in addition to those solicited during the clinical study. Also any "solicited" symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
Time Frame: During the 30-day (Days 0-29) period following each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 149 | 76
Participants | 66 | 19

6. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Diseases (NOCDs) and Medically Significant Conditions
Description: NOCDs assessed include e.g. autoimmune disorders, asthma, type I diabetes. Medically significant AEs assessed include AEs prompting emergency room visits and physician office visits not related to common illnesses or Serious Adverse Events (SAEs) that are not related to common illnesses.
Time Frame: From Day 0 up to Month 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 149 | 76
Participants
  NOCD | 5 | 6
  Medically Significant Conditions | 34 | 10

7. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE)
Description: Serious adverse events assessed include medical occurrences that result in death, is life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 0 up to Month 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 149 | 76
Participants | 2 | 1

8. Secondary Outcome: Number of Subjects With Pregnancies and Their Outcome
Description: Total: the total number of pregnancies in a group. The specific outcomes are also listed.
Time Frame: from Day 0 up to Month 7
Population: Analysis was performed on subjects with a pregnancy.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 0 | 1
Participants
  Total |  | 1
  Elective abortion |  | 1

ADVERSE EVENTS:
Arm/Group | Cervarix Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 2/149 | 1/76
Other Adverse Events (participants affected / at risk) | 144/149 | 70/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=149) | Placebo Group (N=76)
Gastroenteritis viral (Infections and infestations) | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=149) | Placebo Group (N=76)
Upper respiratoy tract infection (Infections and infestations) | 20 | 3
Dysmenorrhea (Reproductive system and breast disorders) | 13 | 3
Headache (Nervous system disorders) | 9 | 4
Injection site pruritus (General disorders) | 9 | 0
Pain (General disorders) | 140 | 64
Redness (General disorders) | 109 | 35
Swelling (General disorders) | 89 | 19
Arthralgia (General disorders) | 35 | 8
Gastrointestinal symptoms (General disorders) | 52 | 16
Headache (General disorders) | 73 | 30
Myalgia (General disorders) | 97 | 33
Rash (General disorders) | 29 | 8
Urticaria (General disorders) | 12 | 2
Fatigue (General disorders) | 103 | 39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.